CLINICAL TRIAL: NCT06903806
Title: Determination of Microbiome Diversity and Inflammation Throughout the GI Tract During Endurance Exercise
Brief Title: Microbiome Sampling During Endurance Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Spencer, Instructor of Medicine, Gastroenterology and Hepatology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-67010
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Exercise-Induced Lactic Acidemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise with microbiome sampling (Experimental): Participants exercise on a treadmill after swallowing a microbiome sampling capsule. They will then repeat this procedure during controlled cooling of body temperature to prevent increased body temperature during exercise.
  Interventions: Other: Treadmill Exercise; Device: Cooling Gloves; Device: Microbiome Capsule

INTERVENTIONS:
Other: Treadmill Exercise — Participants perform moderate to strenuous exercise for up to 20 minutes on a treadmill after swallowing a microbiome sampling capsule.
Device: Cooling Gloves — Cooling gloves to prevent rise in core body temperature during exercise
Device: Microbiome Capsule — Capsule used for collecting intestinal tract contents

SUMMARY:
The small intestine and feces of subjects undergoing endurance exercise will be sampled to examine their microbiome composition

DETAILED DESCRIPTION:
The close relationship between humans and the commensal microbes of their gut microbiota represents vast potential for health maintenance, but most efforts have been focused on disease. Gastrointestinal (GI) problems are very common especially in endurance athletes, and are known to impair performance or subsequent recovery. Moreover, GI symptoms among athletes vary enormously, and some athletes are more prone than others; the links between this variation and the differences in microbiome composition across individuals have not been elucidated. The investigators propose to use a novel, non-invasive sampling technology to quantify the effects of exercise on the GI environment including the small intestines, and aim to establish the potential for dietary interventions to improve recovery from exercise.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

* Males or females 18 years of age or older and 70 years of age or younger at the time of the first Screening Visit.
* ASA Classifications 1 and 2.
* For women of childbearing potential, negative urine pregnancy test within 7 days of Screening Visit. Willingness to use highly effective contraception during the entire study period (e.g.: implants, injectables, oral contraceptives, intra-uterine device or declared abstinence).
* Subject is fluent in English and understands the study protocol and informed consent and is willing and able to comply with study requirements and sign the informed consent form. Non-English speakers will not be included in the study because consent forms are in English, and any instructions during exercise will need to be provided in English.

Exclusion Criteria:

Subjects with any of the following conditions or characteristics must be excluded from the study:

* History of any of the following:
* Prior gastric or esophageal surgery, including lap banding or bariatric surgery
* Bowel obstruction
* Gastric outlet obstruction
* Diverticulitis
* Inflammatory bowel disease
* Ileostomy or colostomy
* Gastric or esophageal cancer
* Achalasia
* Esophageal diverticulum
* Active Dysphagia or Odynophagia
* Active medication use for any gastrointestinal conditions
* Pregnancy or planned pregnancy within 30 days from Screening Visit, or breast-feeding
* Any form of active substance abuse or dependence (including drug or alcohol abuse), unstable medical or psychiatric disorder, or any chronic condition susceptible, in the opinion of the investigator, to interfere with the conduct of the study
* A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the subject while involved in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants completing exercise | 1 day
  Target goal is 80% of subjects will complete their exercise testing

SECONDARY OUTCOMES:
Volume of intestinal fluid from subjects for analysis | 2 weeks
  Target goal is 80% of subjects to have at least 100ul of intestinal fluid collected from microbiome-sampling capsule

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Spencer, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shalon D, Culver RN, Grembi JA, Folz J, Treit PV, Shi H, Rosenberger FA, Dethlefsen L, Meng X, Yaffe E, Aranda-Diaz A, Geyer PE, Mueller-Reif JB, Spencer S, Patterson AD, Triadafilopoulos G, Holmes SP, Mann M, Fiehn O, Relman DA, Huang KC. Profiling the human intestinal environment under physiological conditions. Nature. 2023 May;617(7961):581-591. doi: 10.1038/s41586-023-05989-7. Epub 2023 May 10. PMID 37165188